CLINICAL TRIAL: NCT06047756
Title: Effects of Hippotherapy Versus Swiss Ball Training to Improve Trunk Control and Balance on Spastic Daiplegic Child
Brief Title: Hippotherapy Versus Swiss Ball Training to Improve Trunk Control and Balance on Spastic Daiplegic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/00123Mehrin Wadood
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Cerebral Palsy Spastic Diplegia
MeSH Terms: conditions — Cerebral Palsy | interventions — Equine-Assisted Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hippotherapy (Experimental): Patients suffering with diplegic therapy will perform their exercise protocols on a stationary horse.The child is seat astride the horse wearing a helmet and was encouraged to perform various activities designed to emphasize movement in a forward and upward reaching direction to encourage active postural control, trunk strength, balance and trunk/pelvic dissociation.30 minutes to 1 hour with a frequency ranging from 4 sessions per week and the total duration of horseback riding 6 weeks.
  Interventions: Other: Hippotherapy
- Swiss Ball therapy (Active Comparator): Children of second group will receive swiss ball therapy. Position the child to sit on the ball and giving extension rotation and flexion rotation to the child. This will facilitate trunk rotation by which the upper body is towards the weight bearing hip and away from the weight bearing hip.Training program 4 times per weeks with the treatment session of 30 minutes for 6 weeks duration
  Interventions: Other: Swiss Ball therapy

INTERVENTIONS:
Other: Hippotherapy — Patient will perform different movement of the trunk while sitting on a horse.
  Arms: Hippotherapy
Other: Swiss Ball therapy — Patient will perform movements of trunk on swiss ball
  Arms: Swiss Ball therapy

SUMMARY:
To compare effect in both intervention

DETAILED DESCRIPTION:
In this study we will compare the effects of hippotherapy and swiss ball therapy. Our objectives of the study are To compare the effects of hippotherapy and Swiss ball training, to improve trunk control and balance on spastic diplegic cerebral palsy

ELIGIBILITY:
Inclusion Criteria:• Children (male and female)

* Age group 4 to 11 years
* Subject diagnosed with CP
* Mild Spastic Diaplegic of the lower limbs according to the modified ashworth scale grade 1 to 1+
* GMFM scale sitting balance score less than 20
* Medically stable and able to understand commands

Exclusion Criteria:• Children with mental retardation,

* Epilepsy, other associated neurological disorders, other type of cerebral palsy,
* Attention deficit hyperactivity disorder and sensory issues(poor visual or hearing acuity)

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Gross Motor Functional Scale | 6weeks
  Changes from baseline The Gross Motor Function Measure (GMFM) is an observational clinical tool designed to evaluate change in gross motor function in children with cerebral palsy.Greater score means higher functional level
Trunk Control Measurement Scale | 6 weeks
  Changes from Baseline The TCMS scale assesses seated trunk control in three dimensions. The maximum score is 58 points where 20 points correspond to static balance, 28 to selective movement control, and 10 to the ability to perform dynamic reaching
Pediatric Balance Scale | 6 weeks
  Changes from Baseline Pediatric Balance Scale is a modified version of the Berg Balance Scale that is used to assess functional balance skills in school-aged children. The scale consists of 14 items that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Bashir, MSNMPT, Principal Investigator — Riphah international University Islamabad
Locations (1):
- Helping hand for relief and development, Dīr, Khyberpakhtunkhuwa, Pakistan

IPD SHARING:
Plan to Share IPD: No